CLINICAL TRIAL: NCT01544868
Title: Total Energy Expenditure, Protein Kinetics and Body Composition During Recovery From Severe Burn Injury in Children.
Brief Title: Total Energy Expenditure, Protein Kinetics, and Body Composition in Recovering Burn Children.
Acronym: TEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Kathy Prelack, PhD, RD, Director of Clinical Research, Shriners Hospitals for Children
Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2006P001559
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Energy Expenditure in Burn Children; Protein Turnover in Burn Children
Keywords: Total Energy Expenditure; Protein Balance; Burns
MeSH Terms: conditions — Burns | interventions — Proteolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Energy expenditure measurement (Other): Descriptive measurements
  Interventions: Other: Use of Stable Isotope to Measure Energy Expenditure and Protein Turnover

INTERVENTIONS:
Other: Use of Stable Isotope to Measure Energy Expenditure and Protein Turnover — Two pre-dose urine specimens will be collected prior to an oral dose containing 0.22 g/kg total body water of 100% 18O water (or 1.2 g/kg per body weight of 10% 18O water) and 0.11 g/kg per body weight of 99.9% deuterium oxide. Then the patient will receive a single dose (4mg/kg, less than 2% of normal daily intake of 1.1g per person) of 15N glycine tracer. For this, patients will drink a dose of 15N glycine (4mg.kg 1dissolved in 20 ml of saline) mixed in 50 cc of apple juice or other liquid beverage, followed by a 50 cc wash of water. 24 hour urine collection will commence immediately. Twenty-four hour urines will be used for determining the 15N NH3 and 15N urea enrichment. Each urine container will contain 5 ml of 15N HCl for trapping the urinary ammonium. Urine will be collected each day for 3 days, for determination of the total urinary nitrogen, urea creatinine, and ammonia excretion.

SUMMARY:
The purpose of this study is to measure resting energy expenditure, total energy expenditure, and physical activity in recovering burn children to better understand their relation to impaired growth and nutritional status; and to measure whole body and muscle protein turnover during recovery from burn injury to understand their impact on body composition and energy metabolism. It also aims to look at changes in lean body mass, fat mass, bone mineral density and bone mineral content during rehabilitation and during early convalescence.

DETAILED DESCRIPTION:
Measures of total and resting energy expenditure, protein turnover, body composition and other nutritional and outcome-based measures will be made in patients receiving inpatient rehabilitative care for their burn injury. Patients will consist of acutely burned patients initially admitted to our hospital with burns of 40% of their total body, who have recently recovered from their acute phase of injury and have achieved wound closure as defined by less than 5% open wound area (Group A). In addition, patients admitted to the hospital for "acute rehabilitation", which includes patients in need of rehabilitative therapy will also be included. This latter group (Group B) is unique in that the patients may have open wound areas remaining due to difficulty healing, however are not critically ill. Group B may differ from the typical rehabilitation population seen at our hospital because of their open wounds and because they received care for their initial injury elsewhere. They are included here due to their apparent nutritional compromise and their unique energy and protein requirements that are difficult to predict according to our clinical experience. These patients are most likely to require artificial nutrition support and will benefit from information gained by this study.

Measurements will be made at baseline as defined at the time of wound closure (or at the time of admission for Group B). Subsequent measures will be done as follows: 1) total energy expenditure will be assessed weeks 1-3 and again at weeks 7-9. During weeks 1 and 7, protein turnover studies will take place. Indirect calorimetry and physical activity measures will take place on 2 consecutive days during each week. Lean body mass measurements will be done at the time of wound closure and at discharge. The study will end at the time of discharge.

Resting and total energy expenditure will be done using indirect calorimetry for resting energy expenditure and the doubly labeled water method for total energy expenditure. Briefly, the methodology for doubly labeled water is as follows. Two pre-dose urine specimens will be collected prior to an oral dose containing 0.22 g/kg total body water of 100% 18O water (or 1.2 g/kg per body weight of 10% 18O water) and 0.11 g/kg per body weight of 99.9% deuterium oxide. Three post-dose urine voids will be collected, followed by collection of a morning urine void daily for 7 days. Total energy expenditure by this method will represent the average energy expenditure over a 21-day period. It will be obtained at weeks 1-3 and again at weeks 7-9 weeks during the rehabilitative phase. Resting energy expenditure will be determined using indirect calorimetry by a metabolic cart on 2 consecutive days of each week. Physical activity will be determined by having the patients wear an physical activity monitor (Actical Physical Monitoring System, mini-Mitter, Co., Inc, Bend Oregon) on their wrist, ankle or hand for the entire day twice a week (corresponding to the metabolic cart measurement). This will be worn on 2 days of each week. Protein nutritional status and turnover will be measured using N15 glycine. Three methyl-histidine will be measured at the time of N15 glycine studies (weeks 1 and 7) to assess the contribution of muscle mass to protein turnover. On the day of tracer study, each patient will provide a urine sample, and this urine sample will be collected to determine the basal level of N15 enrichment in urea and ammonia. Then the patient will receive a single dose (4mg/kg, less than 2% of normal daily intake of 1.1g per person) of 15N glycine tracer. For this, patients will drink a dose of 15N glycine (4mg.kg 1dissolved in 20 ml of saline) mixed in 50 cc of apple juice or other liquid beverage, followed by a 50 cc wash of water. 24 hour urine collection will commence immediately. Twenty-four hour urines will be used for determining the 15N NH3 and 15N urea enrichment. Each urine container will contain 5 ml of 15N HCl for trapping the urinary ammonium. Urine will be collected each day for 3 days, for determination of the total urinary nitrogen, urea creatinine, and ammonia excretion.

Lean body mass, fat mass and bone mineral density and content will be determined at baseline (or at the time of wound closure- as is routine care) and at discharge. Body composition components (lean body mass, fat mass and bone mineral density) will be determined for the lumbar spine and the whole body using dual energy x-ray absorptiometry (DXA) with a Discovery QDR 4500 A (Hologic, Waltham, MA) in burned and healthy children. Scanning will be performed by study staff trained and certified in the use of DXA. DXA uses x-ray beams at two photon energies to estimate body composition. Prior to the scan, height will be measured at the time of each measurement session with the subjects standing barefoot and in light clothing using a stadiometer. Measures will be recorded to the nearest 0.5 centimeters respectively. Weight will be taken using a balance scale and recorded to the nearest 0.5 kilograms. DXA measurements will be done by having the patient lie flat on his or her back on the DXA scanning table. Subjects will be positioned by the scanner so that the spine is straight on the table pad. For the lumbar spine measurement, a knee positioner will be placed under the patient's lower legs so that the patient's knees and hip are at a 90 degree angle. To align the C-arm (scanning arm ) of the DXA, a laser line will be positioned 1-2 inches below the patient's ileac crest, centered around the patient's midline. The scan time approximates 10 seconds, exposure is 0.38 mRem. For the whole body scan, the subject will lay on his or her back with their body straight, arms at sides, palms down, separated from thighs. The scanner will rotate the subject's legs inward 25 degrees until the toes touch, using tape around the feet to maintain this position. The subject will be instructed to breathe normally. The total scan time approximates 2.5 to 3.5 minutes with an exposure of 0.26 mRem. Total body fat and lean body mass will be determined by the DEXA as described as part of the whole body bone mineral density scan (only 1 scan session required). Measures of % body fat content and % lean body mass content for the whole body will be obtained using the DEXA software. These values will be compared to age and sex matched pediatric reference data for body composition {{217 Ellis, K.J. 2000; }}.

Because measures of LBM can be confounded by hydration status, a second measure of LBM using bioelectrical impedance will be made at these points and compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 2 less than 18 who have been admitted to our hospital for treatment of an initial wound size of 40% or greater total body surface area burn, which has subsequently healed

Exclusion Criteria:

* hemodynamically unstable
* not receiving enteral nutrition

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Total Energy Expenditure | 4 years
  Tota Energy Expenditure will be determined in this group of burn children

SECONDARY OUTCOMES:
Protein Turnover | 4 years
  Protein synthesis and breakdown will determined by stable isotope methodology

CONTACTS AND LOCATIONS:
Locations (1):
- Shriners Hospitals For Chidren, Boston, Massachusetts, United States